CLINICAL TRIAL: NCT06672861
Title: Development and Validation of the Kansas City Cardiac Dysautonomia Questionnaire (KCDysQ) in Patients With Postural Orthostatic Tachycardia Syndrome, Inappropriate Sinus Tachycardia, and Other Disorders of Cardiac Dysautonomia
Brief Title: Development and Validation of the Kansas City Cardiac Dysautonomia Questionnaire (KCDysQ)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute, Overland Park, KS (Unknown); Midwest Heart and Vascular Specialists, Overland Park, KS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCHRRF-KCDysQ-0014
Record Dates: First submitted 2022-07-06; First posted 2024-11-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Dysautonomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly diagnosed/untreated/incompletely treated for Cardiac Dysautonomia Patients (Other): Newly diagnosed/untreated/incompletely treated for Cardiac Dysautonomia (Postural Orthostatic Tachycardia Syndrome (POTS), Inappropriate Sinus Tachycardia (IST), and Vasovagal syncope (VVS)) Patients
  Interventions: Other: Kansas City Cardiac Dysautonomia Questionnaire (KCDysQ)
- Previously diagnosed/treated/undergone sinus node modification for Cardiac Dysautonomia Patients (Other): Previously diagnosed/treated/previously undergone sinus node modification for Cardiac Dysautonomia Patients (Postural Orthostatic Tachycardia Syndrome (POTS), Inappropriate Sinus Tachycardia (IST), and Vasovagal syncope (VVS)) Patients
  Interventions: Other: Kansas City Cardiac Dysautonomia Questionnaire (KCDysQ)

INTERVENTIONS:
Other: Kansas City Cardiac Dysautonomia Questionnaire (KCDysQ) — To compare in patients with cardiac dysautonomia, newly developed disease specific questionnaire to established generalized SF-36 and EQ-5d questionnaires, as there are no disease specific questionnaires for comparison. These novel and established questionnaires will then be compared among groups who have relatively stable disease or stable symptoms with patients who will be expected to have a change in symptoms and QoL.

SUMMARY:
Main aim will be to compare in patients with cardiac dysautonomia, newly developed disease specific questionnaire to established generalized SF-36 and EQ-5d questionnaires, as there are no disease specific questionnaires for comparison. These novel and established questionnaires will then be compared among groups who have relatively stable disease or stable symptoms with patients who will be expected to have a change in symptoms and QoL.

DETAILED DESCRIPTION:
With the advent of other disease specific questionnaires in patients with cardiac disease such as the AFEQT questionnaire, patients with cardiac dysautonomia have a unique symptom set that can range from mild symptoms to debilitating on a daily scale. Given that they are an underdiagnosed population who often have considerable rates of misdiagnosis, diagnostic delay, and concurrent life limiting factors not addressed by previous QOL assessments, the next logical step therefore is the development and further validation of a QOL questionnaire that serves to respect and represent the 6 domains of QOL as stated by the WHO, with representation of all four health related QOL (HRQoL), as well as focus on underrepresented areas of patients with cardiac dysautonomia.

A novel disease specific KCDysQ questionnaire with questions being gathered from an extensive literature review of QOL measures in this subset of patients as well as interviews and personal interactions with these patients is proposed. It will begin with a 100-item questionnaire and proceed to use a power analysis to further stratify this. For validation of this questionnaire, it is proposed to prospectively recruit all patients with a diagnosis of POTS, IST, or VVS in a single center, and stratify them into patients with a new diagnosis/untreated POTS, IST, or VVS compared with patients who have had symptoms improvement with medication or stable disease who present for routine follow ups. Though an emerging technique and therefore a small but important percentage of this population, patients who have underwent sinus node manipulation for treatment of their IST or POTS as well will also be included, as these subsets of patients have undergone little prior evaluation.

ELIGIBILITY:
Inclusion criteria:

Patients with a Diagnosis of POTS, IST, or vasovagal syncope

Exclusion criteria:

Patients with comorbid chronic conditions causing significant impairments in quality of life, defined as:

* NYHA Class III or IV Heart Failure
* COPD GOLD 3 or 4, Group C or D
* Any patients with current malignancy not in remission
* Any patient with history of Autoimmune disease requiring chronic steroid therapy or immunomodulatory agents: Rheumatoid Arthritis, Lupus, Sarcoidosis, Psoriasis All patients with ESRD requiring hemodialysis All patients with cirrhosis of any origin Any patients with solid organ or bone marrow transplant requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To develop and validate KCDysQ as a quality of life and symptom severity assessment tool | 3 Months
  The primary objective of this study will be to develop and validate KCDysQ as a quality of life and symptom severity assessment tool that can be widely applied to patients with symptoms of cardiac dysautonomia, and doing so by proving the questionnaire's reliability, validity, responsiveness, and acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (3):
- United States (3):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Background] Abed HS, Fulcher JR, Kilborn MJ, Keech AC. Inappropriate sinus tachycardia: focus on ivabradine. Intern Med J. 2016 Aug;46(8):875-83. doi: 10.1111/imj.13093. PMID 27059112
- [Background] Shaw BH, Stiles LE, Bourne K, Green EA, Shibao CA, Okamoto LE, Garland EM, Gamboa A, Diedrich A, Raj V, Sheldon RS, Biaggioni I, Robertson D, Raj SR. The face of postural tachycardia syndrome - insights from a large cross-sectional online community-based survey. J Intern Med. 2019 Oct;286(4):438-448. doi: 10.1111/joim.12895. Epub 2019 Apr 16. PMID 30861229
- [Background] Bagai K, Song Y, Ling JF, Malow B, Black BK, Biaggioni I, Robertson D, Raj SR. Sleep disturbances and diminished quality of life in postural tachycardia syndrome. J Clin Sleep Med. 2011 Apr 15;7(2):204-10. PMID 21509337
- [Background] Benrud-Larson LM, Dewar MS, Sandroni P, Rummans TA, Haythornthwaite JA, Low PA. Quality of life in patients with postural tachycardia syndrome. Mayo Clin Proc. 2002 Jun;77(6):531-7. doi: 10.4065/77.6.531. PMID 12059122
- [Background] Raj SR. Postural tachycardia syndrome (POTS). Circulation. 2013 Jun 11;127(23):2336-42. doi: 10.1161/CIRCULATIONAHA.112.144501. No abstract available. PMID 23753844
- [Background] Ptaszynski P, Kaczmarek K, Ruta J, Klingenheben T, Wranicz JK. Metoprolol succinate vs. ivabradine in the treatment of inappropriate sinus tachycardia in patients unresponsive to previous pharmacological therapy. Europace. 2013 Jan;15(1):116-21. doi: 10.1093/europace/eus204. Epub 2012 Jul 6. PMID 22772053
- [Background] Fedorowski A. Postural orthostatic tachycardia syndrome: clinical presentation, aetiology and management. J Intern Med. 2019 Apr;285(4):352-366. doi: 10.1111/joim.12852. Epub 2018 Nov 23. PMID 30372565
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035